CLINICAL TRIAL: NCT03168776
Title: A Prospective Global Randomized Trial Assessing the Safety and Efficacy of the BuMA Supreme™ Biodegradable Drug Coated Coronary Stent System for Coronary Revascularization in Patients With Stable Coronary Artery Disease or Non-ST Segment Elevation Acute Coronary Syndromes
Brief Title: PIONEER III Trial to Assess Safety and Efficacy of the BuMA Supreme™ Drug Coated Coronary Stent in Patients With Coronary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Collaborators: Nova Vascular LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIN-US-001
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BuMA Supreme Coronary Stent System (Experimental)
  Interventions: Device: BuMA Supreme DES
- Xience or Promus Everolimus Stent System (Active Comparator)
  Interventions: Device: Xience or Promus DES

INTERVENTIONS:
Device: BuMA Supreme DES — Implant BuMA Supreme stent only
  Arms: BuMA Supreme Coronary Stent System
Device: Xience or Promus DES — Implant XIENCE family or Promus family only
  Arms: Xience or Promus Everolimus Stent System

SUMMARY:
The primary objective of this trial is to compare the safety and efficacy of the SINOMED BuMA Supreme biodegradable coronary stent in patients with up to 3 coronary lesions to either the XIENCE or Promus durable polymer coronary stents.

This prospective, global, multi-center, randomized 2:1, single blind study will enroll up to 1632 subjects at up to 130 investigational sites in North America, Japan, and Europe. Subjects will have clinical follow-up in-hospital and at 30 days, 6 months, 12 months, and 2, 3, 4, and 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a male or non-pregnant female ≥20 years of age.
2. The patient has symptomatic ischemic heart disease, including chronic stable angina (and/or objective evidence of myocardial ischemia on functional study or invasive fractional flow reserve [FFR] measurement) or acute coronary syndromes (UA or NSTEMI), that requires elective or urgent percutaneous coronary intervention (PCI).
3. The patient is an acceptable candidate for percutaneous coronary intervention (PCI) with drug-eluting stents, and for emergent coronary bypass graft (CABG) surgery.
4. The patient is willing to comply with specified follow-up evaluations.
5. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has been provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
2. Patients with a history of bleeding diathesis or coagulopathy, contraindications to anti-platelet and/or anticoagulant therapy, or who will refuse transfusion.
3. Patients who are receiving or will require chronic anticoagulation therapy for any reason.
4. Known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, ADP receptor antagonists (clopidogrel, prasugrel, ticagrelor, ticlopidine), cobalt chromium, 316L stainless steel or platinum, sirolimus or its analogues, and/or contrast sensitivity that cannot be adequately pre-medicated.
5. ST-segment elevation myocardial infarction (STEMI) at index presentation or within 7 days prior to randomization.
6. Known LVEF <30% or cardiogenic shock requiring pressors or mechanical circulatory assistance (e.g., intra-aortic balloon pump, left ventricular assist device, other temporary cardiac support blood pump).
7. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation or Cockcroft-Gault formula) or dialysis at the time of screening.
8. Target vessel percutaneous coronary intervention with stent placement in the previous 3 months.
9. Planned elective surgery that would require discontinuation of DAPT within 6 months of the index procedure.
10. Past or pending heart or any other organ transplant, or on the waiting list for any organ transplant.
11. Patients who are receiving immunosuppressant therapy, or who have known immunosuppressive or severe autoimmune disease that will require chronic immunosuppressive therapy. NOTE: Corticosteroid use is permitted.
12. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound data interpretation, or is associated with a life expectancy of less than 1 year.
13. Current participation in another investigational drug or device study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1629 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Study Chair — Center for Interventional Vascular Therapy - Columbia University Medical Center / New York-Presbyterian Hospital, United States; Dean Kereiakes, MD, Principal Investigator — The Christ Hospital Physicians - Ohio Heart & Vascular, United States; Stephan Windecker, MD, Principal Investigator — Bern University Hospital Department for Cardiology, Switzerland; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital, Japan
Locations (58):
- United States (40):
  - Cardiology, PC, Birmingham, Alabama
  - Dignity Health - Mercy Gilbert Medical Center / Chandler Regional Medical Center, Gilbert, Arizona
  - Smidt Heart Institute Cedars-Sinai Maedical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Medstar Washington HWospital Center, Washington D.C., District of Columbia
  - Bethesda Hospital East/Daniel Heart and Vascular Center, Boynton Beach, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - MediQuest Research Group Inc., Ocala, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - St. Vincent's Medical Group, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Northern Michigan Hospital d.b.a. McLaren Northern Michigan, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Essential Health, Duluth, Minnesota
  - North MS Medical Center, Tupelo, Mississippi
  - CHI Health Research Center, Omaha, Nebraska
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Lindner Research Center, Cincinnati, Ohio
  - North Ohio Heart, Elyria, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Genesis Hospital, Zanesville, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Swedish Medical Center, Seattle, Washington
- Belgium (4):
  - Imelda, Bonheiden
  - CHU Charleroi, Charleroi
  - Ziekenhuis Oost Limburg Genk, Genk
  - Jessa Hospital, Hasselt
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Michael's Hospital, Toronto, Ontario
- Shonan Kamakura General Hospital, Kanagawa, Kamakura City, Japan
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - MCL, Leeuwarden
  - Maasstad Ziekenhuis, Rotterdam
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Instituto de Investigación Hospital 12 de Octubre, Madrid
  - Hospital Álvaro Cunqueiro, Vigo
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - University Hospital Geneva HUG, Clinic for Cardiology, Geneva
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lansky AJ, Kereiakes DJ, Baumbach A, Windecker S, Hussain Y, Pietras C, Dressler O, Issever O, Curtis M, Bertolet B, Zidar JP, Smits PC, Alfonso Jimenez Diaz V, McLaurin B, Hofma S, Cequier A, Dib N, Benit E, Mathur A, Brogno D, Berland J, Wykrzykowska J, Piegari G, Brugaletta S, Saito S, Leon MB; PIONEER III Trial Investigators. Novel Supreme Drug-Eluting Stents With Early Synchronized Antiproliferative Drug Delivery to Inhibit Smooth Muscle Cell Proliferation After Drug-Eluting Stents Implantation in Coronary Artery Disease: Results of the PIONEER III Randomized Clinical Trial. Circulation. 2021 Jun;143(22):2143-2154. doi: 10.1161/CIRCULATIONAHA.120.052482. Epub 2021 Apr 6. PMID 33820424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BuMA Supreme Coronary Stent System | Xience or Promus Everolimus Stent System
Started | 1086 | 543
ITT Analysis Population - Sufficient Data to Evaluate Primary Endpoint | 1058 | 530
ITT Completed 12-Month Clinical F/U | 1042 | 522
Completed | 1042 (99.0%) | 522 (99.4%)
Not Completed | 44 | 21

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population excludes 1 subject from the ITT Population who was withdrawn from the study after informed consent but prior to receiving a study device.
Groups:
- BuMA Supreme Coronary Stent System (ITT): The BuMA Supreme Biodegradable Drug Coated Coronary Stent System is a device / drug combination product consisting of a drug-coated balloon expandable stent and a rapid exchange delivery system. The cobalt chromium (CoCr) stent is coated with a very thin, non-erodable layer of poly n-butyl methacrylate (PBMA) that is covalently bonded to the metal surface through a proprietary electro-grafting (eG™) process. A topcoat is then applied that contains sirolimus, the active ingredient, embedded in a biodegradable polymer, poly lactic co-glycolic acid (PLGA).
- Durable Polymer EES (XIENCE or Promus DES) (ITT): The control comparator is durable polymer everolimus-eluting stent systems (DP EES), consisting of the Xience™ family of durable polymer cobalt chromium everolimus-eluting coronary stent systems (Abbott Vascular, Santa Clara, CA, US), and the PROMUS Element™ family of everolimus-eluting coronary stent systems.
- Total: Total of all reporting groups
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT) | Total
Number analyzed (Participants) | 1086 | 542 | 1628
Age, Customized [Count of Participants; unit: Participants]
  Age ≥65 | 567 | 272 | 839
  Age <65 | 519 | 270 | 789
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 148 | 406
  Male | 828 | 394 | 1222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 53 | 144
  Not Hispanic or Latino | 941 | 455 | 1396
  Unknown or Not Reported | 54 | 34 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 129 | 63 | 192
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 34 | 19 | 53
  White | 868 | 427 | 1295
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 53 | 33 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 70 | 36 | 106
  Netherlands | 124 | 62 | 186
  Belgium | 76 | 38 | 114
  United States | 479 | 231 | 710
  Japan | 108 | 55 | 163
  United Kingdom | 45 | 25 | 70
  Switzerland | 11 | 8 | 19
  Spain | 138 | 67 | 205
  France | 35 | 20 | 55
Height [Mean (Standard Deviation); unit: cm] | 171.33 (9.76) | 170.64 (9.92) | 171.10 (9.81)
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 85.68 (19.69) | 85.70 (19.17) | 85.68 (19.52)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 29.06 (5.71) | 29.32 (5.66) | 29.15 (5.69)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 134.1 (22.1) | 133.8 (22.1) | 134.0 (22.1)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 74.9 (12.6) | 75.0 (12.6) | 74.9 (12.6)
Pulse (bpm) [Mean (Standard Deviation); unit: bpm] | 68.9 (12.8) | 69.2 (12.4) | 69.0 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Failure (TLF) and Constituent Elements
Description: TLF is defined as the composite of cardiac death, target vessel related myocardial infarction (TV-MI), and clinically-driven target lesion revascularization (TLR)
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with TLF
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1058 | 530
percentage of subjects with TLF
  TLF | 5.4 [4.1 to 6.9] | 5.1 [3.4 to 7.3]
  Cardiac Death | 0.3 [0.1 to 0.8] | 0.8 [0.2 to 1.9]
  Target vessel MI | 3.4 [2.4 to 4.7] | 4.2 [2.6 to 6.2]
  Clinically Driven TLR | 2.3 [1.5 to 3.4] | 0.9 [0.3 to 2.2]

2. Secondary Outcome: Number of Participants With Cardiac Death
Description: Any death due to proximate cardiac cause (e.g., MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Population: Number of participants with Cardiac Death
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  30 Days | 2 | 1
  6 Months | 3 | 3
  12 Months | 3 | 4
  5 Years | 25 | 16

3. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: All-cause death, myocardial infarction, or target vessel revascularization (reported as a composite)
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  30 Days | 39 | 22
  6 Months | 58 | 33
  12 Months | 79 | 39
  5 Years | 210 | 113

4. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: Defined according to the modified Third Universal Definition as evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia.
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  30 Days | 36 | 21
  6 Months | 43 | 22
  12 Months | 51 | 24
  5 Years | 87 | 47

5. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Definite or probable (ARC-defined), classified as early, late, or very late
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  30 Days | 7 | 2
  6 Months | 7 | 2
  12 Months | 8 | 2
  5 Years | 26 | 14

6. Secondary Outcome: Number of Participants With Bleeding Complications (BARC Definitions)
Description: Evaluated as components and as a composite of BARC Type 3 or 5 bleeding, including:
  Type 3a: Over bleeding plus hemoglobin drop of 3 to <5 g/dL* (provided hemoglobin drop is related to bleed); Any transfusion with over bleeding Type 3b: Overt bleeding plus hemoglobin drop ≥5 g/dL* (provided hemoglobin drop is related to bleed); Cardiac tamponade; Bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid); Bleeding requiring intravenous vasoactive agents Type 3c: Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal); Subcategories confirmed by autopsy or imaging or lumbar puncture; Intraocular bleed comprising vision Type 5: Fatal bleeding
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  30 Days | 8 | 2
  6 Months | 14 | 2
  12 Months | 24 | 5
  5 Years | 44 | 22

7. Secondary Outcome: Lesion Success
Description: Defined as attainment of <30% residual stenosis, as measured by quantitative coronary angiography (QCA) using any percutaneous method [evaluated post-procedure]
Time Frame: Post-Procedure
Measure: Count of Units; unit: Number of Lesions Treated
Units Other Than Participants: Number of Lesions Treated
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Number analyzed (Number of Lesions Treated) | 1275 | 656
Number of Lesions Treated | 1271 | 653

8. Secondary Outcome: Device Success
Description: Defined as attainment of <30% residual stenosis of the target lesion measured by QCA using the assigned device [evaluated post-procedure]
Time Frame: Post-Procedure
Measure: Count of Units; unit: Total Number of Devices
Units Other Than Participants: Total Number of Devices
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Number analyzed (Total Number of Devices) | 1246 | 648
Total Number of Devices | 1212 | 640

9. Secondary Outcome: Procedure Success
Description: Defined as lesion success without the occurrence of in-hospital MACE [evaluated in-hospital]
Time Frame: Post procedure/Prior to Discharge, an average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1074 | 537
Participants | 1042 | 514

10. Secondary Outcome: Clinically-driven Target Vessel Revascularization (TVR)
Description: Any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
  A revascularization is considered clinically driven if angiography at follow-up shows a percent diameter stenosis ≥ 70% (by core lab quantitative coronary angiography assessment) OR percent diameter stenosis ≥ 50% (by core lab quantitative coronary angiography assessment) accompanied by one of the following:103
  1. a positive history of recurrent angina pectoris, presumably related to the target vessel;
  2. objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent) presumably related to the target vessel;
  3. abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve).
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  In-Hospital Prior to Discharge | 2 | 2
  30 Days | 8 | 2
  6 Months | 21 | 11
  12 Months | 38 | 16
  5 years | 98 | 45

11. Secondary Outcome: Target Vessel Failure (TVF)
Description: The composite of cardiac death, target vessel-related myocardial infarction, and clinically-driven target vessel revascularization.
Time Frame: Assessed at 30 days, 6 months, 12 months, and up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
Number analyzed (Participants) | 1086 | 543
Participants
  In-Hospital Prior to Discharge | 26 | 19
  30 Days | 34 | 21
  6 Months | 47 | 30
  12 Months | 66 | 34
  5 Years | 146 | 82

ADVERSE EVENTS:
Time Frame: 5 Years
Description: For all adverse events that represented a potential endpoint event, all relevant medical information (including clinically relevant imaging data, ECG data, and the results of relevant laboratory testing performed as part of the standard of care) was collected and retained as part of the research file to support adverse event analysis and adjudication. Coding by organ class was not performed in this study.
  Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | BuMA Supreme Coronary Stent System (ITT) | Durable Polymer EES (XIENCE or Promus DES) (ITT)
All-Cause Mortality (participants affected / at risk) | 79/1086 | 41/543
Serious Adverse Events (participants affected / at risk) | 210/1086 | 113/543
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BuMA Supreme Coronary Stent System (ITT) (N=1086) | Durable Polymer EES (XIENCE or Promus DES) (ITT) (N=543)
MACE (Cardiac disorders) | 210 (323) | 113 (323) — Major Adverse Cardiac Events (MACE; the composite rate of all-cause death, MI and target vessel revascularization)

LIMITATIONS AND CAVEATS:
The trial did not include all comers, e.g. ST elevation MI, left main disease or chronic total occlusion lesions, therefore, limiting generalizability of results to all patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT03168776/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03168776/SAP_001.pdf